CLINICAL TRIAL: NCT00947778
Title: Analysis of Language and Auditory Abilities in Cochlear Implanted Children: Assessment by an Auditory Learning Programmed Method
Brief Title: Analysis of Language and Auditory Abilities in Cochlear Implanted Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2009-05; 2009-A00343-54
Record Dates: First submitted 2009-07-27; First posted 2009-07-28 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Children With Cochlear Implant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- session of training 1 (Active Comparator): Arm from which members will perform their training session after the first session of evaluation
  Interventions: Other: 3 sessions of evaluation tests; Other: 1 training session
- Session of training 2 (Active Comparator): Arm from which members will perform their training session after the second session of evaluation
  Interventions: Other: 3 sessions of evaluation tests; Other: 1 training session

INTERVENTIONS:
Other: 3 sessions of evaluation tests — 3 sessions of evaluation tests, each session during 15 days
Other: 1 training session — 20 sessions of 30 minutes by week during 24 semaines

SUMMARY:
The cochlear implant appears today as one of the best technique so as to lead the congenital deaf children to speak. However the results in terms of accurate access to language remain partial. These results are usually due to the children own factors (social, educational and handicap ones), one which any action has a limited effect.

Besides, there are external factors on which one can rely : " treatments ". For instance, an early cochlear implant on a child is the main stream to a better access to speak properly later. Another essential point to tackle is the early re-education training which remains essential to the treatment. Yet, there is a gap to fill between the theory and the main assistance in the auditory education practice.

The main objective of this survey is to evaluate the efficiency of this auditory teaching programme (MPAA) over the 4 tested skills (identification, discrimination, the analysis of sounds scenes and its memory) among the pre-speaking cochlear implanted congenital deaf children aged from 4 to 10.

This study will be divided into two phases separated by 3 sessions of evaluation tests.

The first session T1 will occur in the two groups (experimentation on G1 and control on G2), then the first training session will start in group G1.

The second session T2 will occur in the two groups, then the first training session will start in group G2.

The third session T3 will occur in the 2 groups at the end of the experiment.

By training the 4 perceptible operations with different auditory stimulations (speech, music, sounds and electro-acoustic sounds), we are looking for better performance in the trained skills as well as a teaching transfer on other linguistic abilities (phonetics discrimination and speech).

DETAILED DESCRIPTION:
The cochlear implant appears today as one of the best technique so as to lead the congenital deaf children to speak. However the results in terms of accurate access to language remain partial. These results are usually due to the children own factors (social, educational and handicap ones), one which any action has a limited effect.

Besides, there are external factors on which one can rely : " treatments ". For instance, an early cochlear implant on a child is the main stream to a better access to speak properly later. Another essential point to tackle is the early re-education training which remains essential to the treatment. Yet, there is a gap to fill between the theory and the main assistance in the auditory education practice.

Researches on auditory cognitive sciences make the distinctions between different operation treatments ranged from the identification of sounds sources to the discrimination of specific acoustic parameters to the analysis of auditory scenes and the memorization of its sources. (Mc Adams and Bigand, 1994).Each operation implies a specific treatment.

Yet, these operations are not systematically followed by a re-education treatment among deaf children even if one is to know that it has a positive impact on the linguistic skills.

They can be trained by a large range of non linguistic stimuli as these specific stimuli belong to the fundamental auditory cognition, their development lead to benefits on the treatment of all the auditory stimuli. Music is part and parcel of the chosen stimuli, as many critics have proved that music was a source of transfer effect for visual and spatial skills for instance (Giomi-Costa, 2003) A synthesis of these researches has been at the source of the so called " method of programmed auditory skills " whose purpose was to develop the complete auditory skills abilities. This complete teaching programme has been integrated in a playful context for children that allows to control the action, the gesture and the game as well as the sounds atmosphere. This teaching programme is controlled by a computer with a large number of different sounds and which is linked to the playful sphere.

The main objective of this survey is to evaluate the efficiency of this auditory teaching programme (MPAA) over the 4 tested skills (identification, discrimination, the analysis of sounds scenes and its memory) among the pre-speaking cochlear implanted congenital deaf children aged from 4 to 10.

This study will take place in the CHU de La Timone in Marseilles in the ENT children department and is at the heart of a cooperation with Dr Emmanuel Bigand team in Dijon (LEAD CNRS, UMR 5022 à Dijon). The cochlear implant children department in Marseilles gathers a group of more than 70 implanted children aged from 4 to 10 that is in adequacy with the parameters for the method to evaluate.

Two groups of 21 cochlear implant children will be included in this study.

This study will be divided into two phases separated by 3 sessions of evaluation tests.

The first session T1 will occur in the two groups (experimentation on G1 and control on G2), then the first training session will start in group G1.

The second session T2 will occur in the two groups, then the first training session will start in group G2.

The third session T3 will occur in the 2 groups at the end of the experiment.

By training the 4 perceptible operations with different auditory stimulations (speech, music, sounds and electro-acoustic sounds), we are looking for better performance in the trained skills as well as a teaching transfer on other linguistic abilities (phonetics discrimination and speech).

ELIGIBILITY:
Inclusion Criteria:

* children with congenital deaf to speak
* children with cochlear implant Nucleus

Exclusion Criteria:

* children unable to understand orders in the oral or in the language of signs

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2009-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
to evaluate the efficiency of this auditory teaching programme (MPAA) over the 4 tested skills (identification, discrimination, the analysis of sounds scenes and its memory) among the pre-speaking cochlear implanted congenital deaf children. | 18 months

SECONDARY OUTCOMES:
to evaluate the efficiency of this auditory teaching programme (MPAA) over the transfer of learning towards tasks of perception and production of the word | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Roman, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique-Hopitaux de Marseille, Marseille, France